CLINICAL TRIAL: NCT02805517
Title: A Prospective Study of Port Site Pain Following Percutaneous Externally-Assembled Laparoscopic Donor Nephrectomy
Brief Title: Port Site Pain Following Percutaneous Externally-Assembled Laparoscopic Donor Nephrectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Number of kidney donors decreased, not able to enroll subjects at this time
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, D. Duane Baldwin, Professor, Loma Linda University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5160152
Record Dates: First submitted 2016-06-14; First posted 2016-06-20 (Estimated); Results first posted 2022-12-13 (Actual); Last update posted 2022-12-13 (Actual); Status verified 2022-11

CONDITIONS: Laparoscopic Donor Nephrectomy
Keywords: Minimally Invasive Surgical Procedures; Transplant Donors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- PEAL laparoscopic nephrectomy (Experimental): Patients will undergo percutaneous externally-assembled laparoscopic donor nephrectomy using 3 mm instruments.
  Interventions: Device: Percuvance™ Percutaneous Surgical System

INTERVENTIONS:
Device: Percuvance™ Percutaneous Surgical System — Patients will undergo percutaneous externally-assembled laparoscopic donor nephrectomy where one or more 3 mm instruments are added or substituted for conventional 5 or 12 mm trocars.
  Other Names: PERCUTANEOUS EXTERNALLY-ASSEMBLED LAPAROSCOPIC (PEAL)

SUMMARY:
A single-arm prospective internally-controlled study. Patients will undergo Percutaneous Externally-Assembled Laparoscopic (PEAL) donor nephrectomy where one or more 3 mm instruments are added or substituted for conventional 5 or 12 mm trocars. Multiple outcome measures (endpoints) will be measured including time to first opioid use, total inpatient opioid dosage, patient ranking of painfulness of each port site, duration of ileus, time to ambulation, length of hospital stay, presence of any intraoperative or postoperative complications, operating time, estimated blood loss, and other routine parameters collected in a prospective surgical study

DETAILED DESCRIPTION:
Purpose:

Prior investigators have created methods to perform laparoscopic surgeries using smaller instruments and ports in an attempt to improve cosmesis and postoperative pain. However, These methods may be limited by the requirement for smaller instruments with decreased functionality or by the loss of instrument triangulation. We have previously published a study regarding the use of a new surgical paradigm (percutaneous externally assembled laparoscopy, or PEAL) in porcine and cadaveric models in order to allow laparoscopic surgery to take place with improved cosmesis and decreased pain while still allowing the use of larger instruments and maintaining instrument triangulation. We now seek to study the use of these instruments in the human patients undergoing laparoscopic urologic surgery.

The procedures include:

Hundred subjects will be recruited for the study with an expected attrition rate of 10%. Sample size has been minimized, but is necessary for statistical power and conclusions. Subjects will be male and female 18 years or older, of all ethnicities, denominations or other social/economical variations. All participants will speak English fluently in order for consent to be performed properly. Baseline pain score will be calculated through a questionnaire in at the urology clinic.

This is a single-arm prospective internally-controlled study. Patients will undergo percutaneous externally-assembled laparoscopic urologic surgery where one or more 3 mm instruments are added or substituted for conventional 5 or 12 mm trocars. Multiple outcome measures (endpoints) will be measured including time to first opioid use, total inpatient opioid dosage, patient ranking of painfulness of each port site, duration of ileus, time to ambulation, length of hospital stay, presence of any intraoperative or postoperative complications, operating time, estimated blood loss, and other routine parameters collected in a prospective surgical study.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing laparoscopic donor nephrectomy

Exclusion Criteria:

* Patients unwilling to participate in the study
* Patients unfit for laparoscopic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-07-11 (Actual); Primary Completion 2021-05-26 (Actual); Study Completion 2021-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Keheila, MD, Study Director — Loma Linda University Medical Center
Locations (1):
- Loma Linda Medical Center, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arenas JL, Alsyouf M, Jang M, Myklak K, Faaborg D, Khater N, Baldwin DD. Percutaneous Externally Assembled Laparoscopic Instruments: Creation of a New Surgical Paradigm. J Endourol. 2016 Apr;30(4):433-40. doi: 10.1089/end.2015.0240. Epub 2016 Feb 9. PMID 26732739
- [Background] Rossitto C, Gueli Alletti S, Costantini B, Fanfani F, Scambia G. Total Laparoscopic Hysterectomy With Percutaneous (Percuvance) Instruments: New Frontier of Minimally Invasive Gynecological Surgery. J Minim Invasive Gynecol. 2016 Jan;23(1):14-5. doi: 10.1016/j.jmig.2015.09.004. Epub 2015 Sep 18. PMID 26386388
- [Background] Chang J, Boules M, Rodriguez J, Kroh M. Minilaparoscopy with Interchangeable, Full 5-mm End Effectors: First Human Use of a New Minimally Invasive Operating Platform. J Laparoendosc Adv Surg Tech A. 2016 Jan;26(1):1-5. doi: 10.1089/lap.2015.0418. Epub 2015 Nov 30. PMID 26618278

RESULTS

PARTICIPANT FLOW:
Groups:
- PEAL Laparoscopic Nephrectomy: Patients who underwent Percutaneous Externally-Assembled Laparoscopic (PEAL) donor nephrectomy using 3 mm instruments.
  Percuvance™ Percutaneous Surgical System: Patients underwent percutaneous externally-assembled laparoscopic donor nephrectomy where one or more 3 mm instruments were used in addition to conventional 5 or 12 mm trocars and the standard hand-assist port.
Period: Overall Study
Arm/Group | PEAL Laparoscopic Nephrectomy
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- PEAL Laparoscopic Nephrectomy: Patients who underwent percutaneous externally-assembled laparoscopic donor nephrectomy using 3 mm instruments.
  Percuvance™ Percutaneous Surgical System: Patients underwent percutaneous externally-assembled laparoscopic donor nephrectomy where one or more 3 mm instruments were used in addition to conventional 5 or 12 mm trocars and the standard hand-assist port.
Arm/Group | PEAL Laparoscopic Nephrectomy
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Time to First Opioid Use
Description: Measurement of time from leaving the post-anesthesia care unit after surgery until the time of first opioid dispersal, regardless of opioid type.
Time Frame: up to 1 day postoperatively
Population: All patients who underwent percutaneous externally-assembled laparoscopic donor nephrectomy
Measure: Median (Full Range); unit: minutes
Arm/Group | PEAL Laparoscopic Nephrectomy
Number analyzed (Participants) | 6
minutes | 74.5 [28 to 677]

2. Primary Outcome: Total Inpatient Opioid Dosage
Description: Total opioid dosage administered throughout the patient's inpatient stay. Measured in units of Morphine Milligram Equivalents (MME).
Time Frame: 3 days postoperatively
Population: Patients who underwent percutaneous externally-assembled laparoscopic donor nephrectomy
Measure: Mean (Standard Deviation); unit: Morphine Milligram Equivalents (MME)
Groups:
- PEAL Laparoscopic Nephrectomy: Patients who underwent percutaneous externally-assembled laparoscopic donor nephrectomy using 3 mm instruments.
  Percuvance™ Percutaneous Surgical System: Patients will undergo percutaneous externally-assembled laparoscopic donor nephrectomy where one or more 3 mm instruments are added or substituted for conventional 5 or 12 mm trocars.
Arm/Group | PEAL Laparoscopic Nephrectomy
Number analyzed (Participants) | 6
Morphine Milligram Equivalents (MME) | 31.3 (9.3)

3. Primary Outcome: Pain Score of All Surgical Sites
Description: A patient-reported pain score (on a scale of 1-10, with 10 being the worst) for each of the four port-site incisions, as measured by the Brief Pain Inventory. Scores were measured on both post-operative day one and on post-operative day two. The four port-site incisions which patients ranked pain scores for were: #1 - Hand-assist Port; #2 - 12 mm Port; #3 - 5 mm Port; #4 - Percutaneous Externally-Assembled Laparoscopic (PEAL) Port. A mean pain score was calculated by averaging the data across the two days.
Time Frame: up to 2 days postoperatively
Population: Patients who underwent percutaneous externally-assembled laparoscopic donor nephrectomy
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Hand-assist Port-site Location: Patient reported scores of the hand-assist port-site pain level. Mean of both post-operative days one and two. All patients had one hand-assist port.
- 12 mm Trochar Port-site Location: Patient reported scores of the 12mm port-site pain level. Mean of both post-operative days one and two. All patients had one 12mm port.
- 5 mm Trochar Port-site Location: Patient reported scores of the 5 mm port-site pain level. Mean of both post-operative days one and two. All patients had one 5 mm port.
- Percutaneous Externally Assembled Laparoscopic (3 mm) Port-site Location: Patient reported scores of the Percutaneous Externally Assembled Laparoscopic (3 mm) port-site pain level. Mean of both post-operative days one and two. All patients had one Percutaneous Externally Assembled Laparoscopic (3 mm) port.
Arm/Group | Hand-assist Port-site Location | 12 mm Trochar Port-site Location | 5 mm Trochar Port-site Location | Percutaneous Externally Assembled Laparoscopic (3 mm) Port-site Location
Number analyzed (Participants) | 3 | 3 | 3 | 3
score on a scale | 5.6 (2.1) | 5.4 (1.9) | 5.2 (2.6) | 2.2 (1.7)

4. Secondary Outcome: Post-operative Ileus
Description: Duration of post-operative ileus as measured by days until return of normal bowel function was noted.
Time Frame: up to 3 days post-operatively
Population: Patients who underwent donor nephrectomy
Measure: Median (Full Range); unit: days
Arm/Group | PEAL Laparoscopic Nephrectomy
Number analyzed (Participants) | 6
days | 2 [1 to 3]

5. Secondary Outcome: Time to Ambulation
Description: Number of post-operative days before patient was noted to be ambulating.
Time Frame: 3 days post-operatively
Population: Patients who underwent donor nephrectomy
Measure: Median (Full Range); unit: days
Arm/Group | PEAL Laparoscopic Nephrectomy
Number analyzed (Participants) | 6
days | 1.5 [1 to 3]

6. Secondary Outcome: Length of Hospital Stay
Description: Number of days admitted to the hospital from surgery until hospital discharge
Time Frame: up do 4 days post-operatively
Population: Patients who underwent donor nephrectomy
Measure: Mean (Standard Deviation); unit: days
Arm/Group | PEAL Laparoscopic Nephrectomy
Number analyzed (Participants) | 6
days | 2.23 (0.59)

7. Secondary Outcome: Presence of Intraoperative Complications
Description: The number of patients with an intraoperative complication.
Time Frame: Intraoperatively
Population: Patients who underwent donor nephrectomy
Measure: Count of Participants; unit: Participants
Arm/Group | PEAL Laparoscopic Nephrectomy
Number analyzed (Participants) | 6
Participants | 0

8. Secondary Outcome: Length of Operative Time
Description: Duration of surgical operation from incision time to procedure stop time
Time Frame: Intraoperatively (up to 6 hours)
Population: Patients who underwent donor nephrectomy
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | PEAL Laparoscopic Nephrectomy
Number analyzed (Participants) | 6
hours | 3.4 (0.3)

9. Secondary Outcome: Estimated Intraoperative Blood Loss
Description: Estimated Blood Loss during the nephrectomy procedure
Time Frame: Intraoperatively (up to 6 hours)
Population: Patients who underwent donor nephrectomy
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | PEAL Laparoscopic Nephrectomy
Number analyzed (Participants) | 6
mL | 33.3 (11.8)

ADVERSE EVENTS:
Time Frame: Up to patients' second clinical follow-up visit, occurring at approximately the six month mark.
Description: Not different from clinicaltrials.gov definitions
Arm/Group | PEAL Laparoscopic Nephrectomy
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PEAL Laparoscopic Nephrectomy (N=6)
Post-operative nausea (Gastrointestinal disorders) | 1 (1) — Self-limited post-operative nausea
Post-operative dizziness (Nervous system disorders) | 1 (1) — Self-limited post-operative dizziness

LIMITATIONS AND CAVEATS:
Although this was a prospective single-blinded study, it was limited by a modest sample size as the performance of donor nephrectomy surgeries transitioned to a separate surgical department not participating in this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-05-03): https://cdn.clinicaltrials.gov/large-docs/17/NCT02805517/Prot_000.pdf
  • Informed Consent Form (2016-06-24): https://cdn.clinicaltrials.gov/large-docs/17/NCT02805517/ICF_001.pdf